CLINICAL TRIAL: NCT01390363
Title: Adolescent Immunization Recall Systems: A Randomized Controlled Trial
Brief Title: Study of Adolescent Immunization Recall Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Kathryn S. Brigham, Fellow, Boston Children's Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 10-01-0025
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Immunization; Reminder Systems
Keywords: immunization; reminder systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- control (No Intervention): This study arm will receive usual clinical care, but no specific intervention will be made to inform the parent or adolescent that the adolescents is overdue for a routine vaccine.
- Parent Only Group (Experimental): Parent Only Phone Call
  Interventions: Other: Parent Only Phone Call
- Parent and Adolescent Group (Experimental): Parent and Adolescent Phone Call
  Interventions: Other: Parent and Adolescent Phone Call

INTERVENTIONS:
Other: Parent Only Phone Call — A telephone call will be made to the parent/guardian informing them that the adolescent has not received one or more vaccines (Td/Tdap in the past 5 years, the MCV4 vaccine, or the 2nd VZV vaccine). The phone call will include a brief informational statement about the vaccine(s) that the adolescent has not yet received. Up to 4 telephone calls will be attempted. As part of the phone call, we will offer to schedule an appointment for the adolescent to receive the missing immunization(s). We will also ask them to mail or fax to the Adolescent/Young Adult Medicine clinic records of immunizations given at other sites.
  Arms: Parent Only Group
Other: Parent and Adolescent Phone Call — A telephone call will be made to the parent/guardian informing them that the adolescent has not received one or more vaccines (Td/Tdap in the past 5 years, the MCV4 vaccine, or the 2nd VZV vaccine). The phone call will include a brief informational statement about the vaccine(s) that the adolescent has not yet received. Up to 4 telephone calls will be attempted. As part of the phone call, we will offer to schedule an appointment for the adolescent to receive the missing immunization(s). We will also ask them to mail or fax to the Adolescent/Young Adult Medicine clinic records of immunizations given at other sites. We will also ask permission to speak with the adolescent as well, and if granted, will make up to 4 phone calls to the adolescent to convey the same message.
  Arms: Parent and Adolescent Group

SUMMARY:
The purpose of this study is to determine whether contacting the parents of adolescents overdue for routine vaccines or contacting both the parents AND adolescents overdue to routine vaccines improves immunization rates as compared to usual care.

DETAILED DESCRIPTION:
This randomized controlled trial is a 3-armed study designed to evaluate an immunization recall system in adolescents. In the control arm (Group 1), the adolescents will receive usual care, in which they will primarily receive immunizations at annual physical exams, or as recommended by providers at urgent care visits. In one intervention arm (Group 2), the parent/guardian will receive a telephone call informing them that the adolescent is overdue for one or more immunizations (conjugated Neisseria meningitidis (MCV4) vaccine, tetanus-diphtheria-pertussis (Tdap) booster, and/or the second varicella (VZV) vaccine). In the second intervention arm (Group 3), both the parent/guardian and the adolescent will receive a telephone call informing them that the adolescent is overdue for one or more immunizations. Immunization rates will be compared between the 3 groups at a four week and a twelve month follow up period.

ELIGIBILITY:
Inclusion Criteria:

* at least 13 years of age and under 18 years of age
* had a billing code for an annual physical exam in the past 3 years at the Adolescent/Young Adult Medical Practice at Children's Hospital Boston
* immunization record shows one of the following: no tetanus containing vaccine in the previous 5 years; no MCV4 vaccine; and/or has received the 1st VZV vaccine but not the 2nd VZV vaccine and has no documented history of the chicken pox

Exclusion Criteria:

* immunization record shows no vaccines or only influenza vaccines
* sibling enrolled in the study
* in the custody of the Department of Youth Services
* in the custody of the Department of Child and Family Services

Ages: 13 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 420 (Actual)
Dates: Start 2010-05-01 (Actual); Primary Completion 2011-07-31 (Actual); Study Completion 2011-07-31 (Actual)

PRIMARY OUTCOMES:
receipt of vaccine of interest at 28 days | 28 days
  Vaccination records are assessed 28 days after the intervention to see if Tdap, MCV4, or the 2nd VZV vaccine were administered.

SECONDARY OUTCOMES:
receipt of vaccine of interest at 1 year | 1 year
  Immunization records are assessed 1 year after the intervention to assess for receipt of Tdap, MCV4, and/or the 2nd VZV vaccine.
receipt of other vaccines at 28 days | 28 days
  Immunization records are assessed 28 days after the intervention to assess for receipt of any vaccine other than Tdap, MCV4, and the 2nd VZV.
receipt of other vaccines at 1 year | 1 year
  Immunization records are assessed 1 year after the intervention to assess for receipt of any vaccine other than Tdap, MCV4, and the 2nd VZV.
receipt of prior vaccines at 28 days | 28 days
  We will assess the immunization record at 28 days to see if it has been updated with vaccines given prior to the enrollment date to see if we successfully obtained copies of immunization records at other healthcare sites.
receipt of prior vaccines at 1 year | 1 year
  We will assess the immunization record at 1 year to see if it has been updated with vaccines given prior to the enrollment date to see if we successfully obtained copies of immunization records at other healthcare sites.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn S Brigham, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Brigham KS, Woods ER, Steltz SK, Sandora TJ, Blood EA. Randomized controlled trial of an immunization recall intervention for adolescents. Pediatrics. 2012 Sep;130(3):507-14. doi: 10.1542/peds.2012-0471. Epub 2012 Aug 20. PMID 22908112